CLINICAL TRIAL: NCT05180266
Title: The Effect of Therapeutic Touch and Music Listening on Sleep Quality, Menopausal Symptoms and Quality of Life in Menopausal Women
Brief Title: Therapeutic Touch and Music in The Menopausal Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Fatma Keskin, Research Assistant, Inonu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: menopause
Record Dates: First submitted 2021-11-28; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Menopause
Keywords: Menopausal Symptoms; Sleep Quality; Therapeutic Touch; Music listening
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Intervention Model Description: After the preliminary test is applied to the experimental groups, therapeutic touch will be applied to one group by the researcher and music listening will be applied to the other group.
  Once a week for four weeks after the preliminary test data Therapeutic Touch Group; Therapeutic Touch application will be performed by the researcher at the appointed time. Each therapeutic touch will take 15 minutes, in accordance with the literature information. At the end of the fourth week, the final test data will be obtained.
  Music Listening Group: After the preliminary test data, women will be asked to listen to relaxation music every day for four weeks for 30 minutes before bedtime in a comfortable environment at home. At the end of the fourth week, the final test data will be obtained.
  To the Control Group; no intervention will be made to women after the preliminary test data.At the end of the fourth week, the final test data will be obtained.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapeutic Touch Group (Experimental): In order to examine the effects of therapeutic touch on menopausal symptoms, sleep and quality of life, women will be given therapeutic touch for 15 minutes, once a week for four weeks.Therapeutic touchis a form of descriptive treatment that lasts approximately 15-20 minutes, in which hands are used on or near the body to correct abnormalities in the person's energy field and to achieve healing, and the energy in the universe is transferred from the practitioner's hands to the applied individual.
  Interventions: Other: Therapeutic Touch
- Music Listening Group (Experimental): The women were asked to listen to the relaxation music included in the relaxation exercises CD prepared by the Turkish Psychological Association every day for four weeks in a comfortable environment at home for 30 minutes before bedtime.
  Interventions: Other: Music Listening Group
- Control Group (Other): No action will be taken on the control group for four weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Therapeutic Touch — Each of the women will be informed about the purpose and content of the study at the first meeting, and informed consent will be obtained from the women who meet the conditions for participation and agree to participate. The pre-test data in the research will be obtained with the Participant Identification Form, PSQI,MRS and MENQOL. After pre-test data collection, women will be given an appointment for therapeutic administration.The therapeutic touch group will be applied to the therapeutic touch group once a week for four weeks in a suitable room in the Faculty of Nursing and on the specified day and time by the researcher.At the end of the fourth week, post-test data will be obtained by filling in PSQI, MRS and MENQOL again.
  Arms: Therapeutic Touch Group
Other: Music Listening Group — Each of the women was informed about the purpose and content of the study at the first meeting, and informed consent was obtained from the women who met the conditions for participation and accepted to participate.The pre-test data in the research will be obtained with the Participant Identification Form, PSQI, MRS and MENQOL. Music stream, music will be uploaded to mobile phones. He will be asked to listen to music (relaxation music in the relaxation exercises CD prepared by the Turkish Psychological Association) for 30 minutes before going to sleep every day for four weeks. At the end of the fourth week, post-test data will be obtained by filling in PSQI, MRS and MENQOL again
  Arms: Music Listening Group
Other: Control Group — Each of the women will be informed about the purpose and content of the study at the first meeting, and informed consent will be obtained from the women who meet the conditions for participation and agree to participate.The pre-test data in the research will be obtained with the Participant Identification Form, PSQI, MRS and MENQOL. No action will be taken on the control group for four weeks. At the end of the fourth week, post-test data will be obtained by filling in PSQI, MRS and MENQOL again.
  Arms: Control Group

SUMMARY:
Menopause is a natural phenomenon and physiological process in middle-aged women. It is noted that women most often complain of vasomotor symptoms and sleep disorders during the menopausal period, and therefore their quality of daily life is negatively affected. Reduce symptoms and improve quality of life for menopausal women they are applying for medical approaches due to the side effects of the method compared to music, yoga, aromatherapy, therapeutic massage, physical exercise, sleep hygiene education, therapeutic touch, acupressure, acupuncture and cognitive behavioral therapy as a non pharmacological methods, it is observed that they resort to such methods. Therefore, the aim of this study is to investigate the effect of therapeutic touch and music listening on sleep quality, menopausal symptoms and quality of life in menopausal women. Therefore, the aim of this study is to investigate the effect of therapeutic touch and music listening on sleep quality, menopausal symptoms and quality of life in menopausal women.

DETAILED DESCRIPTION:
Menopause is a long period of life characterized by the permanent termination of the menstrual cycle due to the cessation of ovarian functions. It is the most important midlife crisis in which special physical and psychological differences occur, often associated with a decrease in estrogen levels. Although the natural age of menopause varies, it usually ranges from 40 to 58 years, and the average age of menopause is accepted as 51. When the average life expectancy of women is accepted as 80 years, women spend about a third or more of their life in the postmenopausal period.

Along with the decrease in estrogen during menopause, symptoms related to hot flashes, night sweats, palpitations, irritability and sleep disorders are common. Especially sleep disorders are higher than in the premenopausal period. It has been reported that approximately 40-60% of menopausal women have sleep-related symptoms with night awakenings as the most common complaint. In the study of Lima et al. in which they included 819 climacteric women in Brazil; Deterioration in sleep quality was detected in 67% of the sample, more prominently in postmenopausal women. The most common complaints during menopause are deterioration of sleep quality and chronic insomnia. Untreated sleep disorders and menopausal symptoms adversely affect health and especially reduce quality of life. When the literature is examined, poor sleep quality and insufficient sleep duration; hormonal changes, poor physical health, obesity, cardiovascular disease, diabetes, irritability, physical and mental burnout, and poor quality of life, such as short-term and long-term outcomes. It is stated that the symptoms seen in the menopausal period negatively affect the quality of life of women.

Although the effective treatment to be used to solve the sleep problems experienced during the menopause period, reduce the menopausal symptoms and improve the quality of life is medication or hormonal therapy, the use of non-pharmacological methods is increasing due to the potential side effects of these treatments and the harm outweighing the benefit. Some of these methods are music, yoga, aromatherapy, therapeutic massage, physical exercise, sleep hygiene education, therapeutic touch, acupressure, acupuncture and cognitive behavioral therapy methods.

Therapeutic touch, which is among the non-pharmacological methods that have started to be preferred in recent years, is the interpretation of an ancient healing experience in the modern age. It is a non-invasive nursing intervention that channels energy using the hands. There are no known side effects associated with the use of therapeutic touch. Therapeutic touch is beneficial in reducing anxiety, pain and depression, and increasing relaxation and well-being.Therefore, this calming effect of therapeutic touch also facilitates falling asleep and can improve quality of life by easing menopausal symptoms. Another widely used non-pharmacological method is recital. Perceived calming music lowers catecholamine levels, respiratory rate, heart rate, and blood pressure. Therefore, by roviding physiological and psychological relaxation, music helps individuals to sleep better, reduce menopausal symptoms, and improve quality of life. In a meta analysis study, it was determined that listening to calming music effectively improved sleep quality.

When the literature was examined, no study was found that examined the effects of therapeutic touch and music listening on sleep quality, menopausal symptoms and menopausal quality of life in menopausal women. It is thought that the findings obtained from the research will contribute to the literature. Based on all these, the aim of this study is to examine the effects of therapeutic touch and music listening on sleep quality, menopausal symptoms and quality of life in menopausal women.

Purpose Of The Study The aim of the study was to investigate the effect of therapeutic touch and music listening on sleep quality, menopausal symptoms and quality of life in menopausal women.

Research Hypotheses H10: Therapeutic touch does not affect sleep quality in menopausal women H11: Therapeutic touch affects sleep quality in menopausal women H20: Therapeutic touch does not affect menopausal symptoms in menopausal women H21: Therapeutic touch affects menopausal symptoms in menopausal women H30: Therapeutic touch does not affect quality of life in menopausal women H31: Therapeutic touch affects quality of life in menopausal women H40: Music listening does not affect sleep quality in menopausal women H41: Listening to music affects sleep quality in menopausal women H50: Listening to music does not affect menopausal symptoms in menopausal women H51: Listening to music affects menopausal symptoms in menopausal women H60: Music listening does not affect quality of life in menopausal women H61: Music listening affects quality of life in menopausal women

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 45-59
* Not taking Hormone Replacement Therapy,
* No psychiatric history,
* Women who do not use any other CAM methods will be included in the study.

Exclusion Criteria:

* Those who are in surgical menopause,
* Having auditory problems that prevent listening to music,
* Using any other TAT method,
* Women who use drugs that affect sleep (using antidepressant, antihistamine, benzodiazepan, hypnotic and narcotic drugs) will be excluded from the study.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-08-25 (Estimated); Study Completion 2022-08-25 (Estimated)

PRIMARY OUTCOMES:
The effect of therapeutic touch on sleep quality | eleven months
  Pittsburgh Sleep Quality Index: The index consists of a total of 24 questions and 7 components. The sum of the scores from the seven components gives the total Pittsburgh Sleep Quality Index score. The total Pittsburgh Sleep Quality Index score can take a value between 0-21. The sleep quality of individuals with a total Pittsburgh Sleep Quality Index score of 5 or less was "good"; The sleep quality of individuals with a score above 5 points is evaluated as "poor".
  Pre-test data in the research will be obtained with the Menopause Symptoms Rating Scale. After completing the scale, women will receive therapeutic touch once a week for four weeks. At the end of the fourth week, the Menopause Symptoms Rating Scale will be filled again.
The effect of therapeutic touch on menopausal symptoms | eleven months
  Menopause Symptoms Rating Scale : There are a total of 11 questions on the Likert-type scale, including menopausal complaints. Each question is scored from 0 to 4. While the minimum score that can be taken from the scale is 0, the maximum score is 44. The increase in the total score obtained from the scale shows the increase in the severity of the complaints, while at the same time it shows that the quality of life is negatively affected.
  Pre-test data in the research will be obtained with the Menopause Symptoms Rating Scale. After completing the scale, women will receive therapeutic touch once a week for four weeks. At the end of the fourth week, the Menopause Symptoms Rating Scale will be filled again.
The effect of therapeutic touch on quality of life | eleven months
  Menopause-Specific Quality of Life Scale: The validity and reliability of the scale was determined by Kharbouch and Şahin in 2007 by adapting the scale to Turkish society Menopause-Specific Quality of Life Scale is a 29-item Likert-type scale. Each question score is ranked from 0 to 6. A score of 0 indicates that women do not have any problems with that subject. A score of 1 indicates that there is a problem with that subject, it is experienced, but it is not disturbing at all. Scores between 2 and 6 indicate the severity and increasing degrees of the existing problem. An increase in the scale score indicates an increase in the severity of the complaints.
  Pre-test data in the research will be obtained with the Menopause Specific Quality of Life Scale. After completing the scale, women will receive therapeutic touch once a week for four weeks. At the end of the fourth week, the Menopause-Specific quality of life scale will be filled again.
The effect of listening to music on sleep quality | eleven months
  Pittsburgh Sleep Quality Index: The index consists of a total of 24 questions and 7 components. The sum of the scores from the seven components gives the total Pittsburgh Sleep Quality Index score. The total Pittsburgh Sleep Quality Index score can take a value between 0-21. The sleep quality of individuals with a total Pittsburgh Sleep Quality Index score of 5 or less was "good"; The sleep quality of individuals with a score above 5 points is evaluated as "poor".
  Pre-test data in the study will be obtained with the Pittsburgh Sleep Quality Index. After the scale is filled, relaxation music will be sent to the women's phones. He will be asked to listen to this music for 30 minutes before going to sleep for four weeks. At the end of the fourth week, the Pittsburgh Sleep Quality Index will be administered again.
The effect of listening to music on menopausal symptoms | eleven months
  Menopause Symptoms Rating Scale : The Turkish validity and reliability study of the scale was carried out by Gürkan in 2005. There are a total of 11 questions on the Likert-type scale, including menopausal complaints. Each question is scored from 0 to 4. While the minimum score that can be taken from the scale is 0, the maximum score is 44. The increase in the total score obtained from the scale shows the increase in the severity of the complaints, while at the same time it shows that the quality of life is negatively affected.
  Pre-test data in the study will be obtained with the Menopause Symptoms Rating Scale. After the scale is filled, relaxation music will be sent to the women's phones. He will be asked to listen to this music for 30 minutes before going to sleep for four weeks. At the end of the fourth week, the Menopause Symptoms Rating Scale will be administered again.
The effect of listening to music on quality of life | eleven months
  Menopause-Specific Quality of Life Scale: Menopause-Specific Quality of Life Scale is a 29-item Likert-type scale. Each question score is ranked from 0 to 6. A score of 0 indicates that women do not have any problems with that subject. A score of 1 indicates that there is a problem with that subject, it is experienced, but it is not disturbing at all. Scores between 2 and 6 indicate the severity and increasing degrees of the existing problem. An increase in the scale score indicates an increase in the severity of the complaints.
  Pre-test data in the study will be obtained with the Menopause-Specific Quality of Life Scale. After the scale is filled, relaxation music will be sent to the women's phones. He will be asked to listen to this music for 30 minutes before going to sleep for four weeks. At the end of the fourth week, the Menopause-Specific Quality of Life Scale will be administered again.

CONTACTS AND LOCATIONS:
Overall Officials: FATMA KESKİN, Principal Investigator — Inonu University; YURDAGÜL YAĞMUR, Professor, Study Director — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abedian Z, Eskandari L, Abdi H, Ebrahimzadeh S. The Effect of Acupressure on Sleep Quality in Menopausal Women: A Randomized Control Trial. Iran J Med Sci. 2015 Jul;40(4):328-34. PMID 26170519
- [Background] Marlatt KL, Beyl RA, Redman LM. A qualitative assessment of health behaviors and experiences during menopause: A cross-sectional, observational study. Maturitas. 2018 Oct;116:36-42. doi: 10.1016/j.maturitas.2018.07.014. Epub 2018 Jul 21. PMID 30244777
- [Background] Kamalifard M, Farshbaf-Khalili A, Namadian M, Ranjbar Y, Herizchi S. Comparison of the effect of lavender and bitter orange on sleep quality in postmenopausal women: A triple-blind, randomized, controlled clinical trial. Women Health. 2018 Sep;58(8):851-865. doi: 10.1080/03630242.2017.1353575. Epub 2017 Aug 25. PMID 28749734
- [Background] Adimi Naghan P, Hassani S, Sadr M, Malekmohammad M, Khoundabi B, Setareh J, Seyedmehdi SM, Seifi S. Sleep Disorders and Mental Health in Menopausal Women in Tehran. Tanaffos. 2020 Jan;19(1):31-37. PMID 33101429
- [Background] Xu Q, Lang CP. Examining the relationship between subjective sleep disturbance and menopause: a systematic review and meta-analysis. Menopause. 2014 Dec;21(12):1301-18. doi: 10.1097/GME.0000000000000240. PMID 24800878
- [Background] Moudi A, Dashtgard A, Salehiniya H, Sadat Katebi M, Reza Razmara M, Reza Jani M. The relationship between health-promoting lifestyle and sleep quality in postmenopausal women. Biomedicine (Taipei). 2018 Jun;8(2):11. doi: 10.1051/bmdcn/2018080211. Epub 2018 May 28. PMID 29806589
- [Background] Cintron D, Lipford M, Larrea-Mantilla L, Spencer-Bonilla G, Lloyd R, Gionfriddo MR, Gunjal S, Farrell AM, Miller VM, Murad MH. Efficacy of menopausal hormone therapy on sleep quality: systematic review and meta-analysis. Endocrine. 2017 Mar;55(3):702-711. doi: 10.1007/s12020-016-1072-9. Epub 2016 Aug 11. PMID 27515805
- [Background] Cao Y, Yin X, Soto-Aguilar F, Liu Y, Yin P, Wu J, Zhu B, Li W, Lao L, Xu S. Effect of acupuncture on insomnia following stroke: study protocol for a randomized controlled trial. Trials. 2016 Nov 16;17(1):546. doi: 10.1186/s13063-016-1670-0. PMID 27852282
- [Background] Lima AM, Rocha JSB, Reis VMCP, Silveira MF, Caldeira AP, Freitas RF, Popoff DAV. [Loss of quality of sleep and associated factors among menopausal women]. Cien Saude Colet. 2019 Jul 22;24(7):2667-2678. doi: 10.1590/1413-81232018247.19522017. Portuguese. PMID 31340284
- [Background] Attarian H, Hachul H, Guttuso T, Phillips B. Treatment of chronic insomnia disorder in menopause: evaluation of literature. Menopause. 2015 Jun;22(6):674-84. doi: 10.1097/GME.0000000000000348. PMID 25349958
- [Background] Crivello, A., Barsocchi, P., Girolami, M., & Palumbo, F. (2019). The meaning of sleep quality: a survey of available technologies. IEEE access, 7, 167374-167390.
- [Background] Troynikov O, Watson CG, Nawaz N. Sleep environments and sleep physiology: A review. J Therm Biol. 2018 Dec;78:192-203. doi: 10.1016/j.jtherbio.2018.09.012. Epub 2018 Oct 5. PMID 30509635
- [Background] Hachul, H., & Polesel, D. N. (2017). Insomnia pharmacotherapy: a review of current treatment options for insomnia in menopause. Current sleep medicine reports, 3(4), 299-305.
- [Background] Afonso RF, Hachul H, Kozasa EH, Oliveira Dde S, Goto V, Rodrigues D, Tufik S, Leite JR. Yoga decreases insomnia in postmenopausal women: a randomized clinical trial. Menopause. 2012 Feb;19(2):186-93. doi: 10.1097/gme.0b013e318228225f. PMID 22048261
- [Background] Johnson A, Roberts L, Elkins G. Complementary and Alternative Medicine for Menopause. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X19829380. doi: 10.1177/2515690X19829380. PMID 30868921
- [Background] HÖzcan, H., Çakmak, S., & Salman, E. (2020). Complementary and Alternative Medicine Methods Used for Sleep Disturbance in Menopause. Journal of Turkish Sleep Medicine, 3, 207-213.
- [Background] Vardar, O., Özkan, S., & Sercekus, P. (2020). Postmenopozal kadınlarda uygulanan egzersiz programının uyku kalitesine etkisi. Cukurova Medical Journal, 45(3), 1108-1114.
- [Background] j. V. Dall, "Promoting sleep with therapeutic touch," Addict. Nurs. Netw., vol. 5, no. 1, pp. 23-24, 1993.
- [Background] Tabatabaee A, Tafreshi MZ, Rassouli M, Aledavood SA, AlaviMajd H, Farahmand SK. Effect of Therapeutic Touch in Patients with Cancer: a Literature Review. Med Arch. 2016 Apr;70(2):142-7. doi: 10.5455/medarh.2016.70.142-147. Epub 2016 Apr 1. PMID 27194823
- [Background] Cordi MJ, Ackermann S, Rasch B. Effects of Relaxing Music on Healthy Sleep. Sci Rep. 2019 Jun 24;9(1):9079. doi: 10.1038/s41598-019-45608-y. PMID 31235748
- [Background] Liu YH, Lee CS, Yu CH, Chen CH. Effects of music listening on stress, anxiety, and sleep quality for sleep-disturbed pregnant women. Women Health. 2016;56(3):296-311. doi: 10.1080/03630242.2015.1088116. Epub 2015 Sep 11. PMID 26361642
- [Background] Dickson GT, Schubert E. How does music aid sleep? literature review. Sleep Med. 2019 Nov;63:142-150. doi: 10.1016/j.sleep.2019.05.016. Epub 2019 Jun 8. PMID 31655374
- [Background] Chen CT, Tung HH, Fang CJ, Wang JL, Ko NY, Chang YJ, Chen YC. Effect of music therapy on improving sleep quality in older adults: A systematic review and meta-analysis. J Am Geriatr Soc. 2021 Jul;69(7):1925-1932. doi: 10.1111/jgs.17149. Epub 2021 Apr 20. PMID 33880759
- [Background] J. Cohen, Statistical Power Analysis for the Behavioral Sciences., 2nd ed. 1988.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] M. Ağargün, H. Kara, and Ö. Anlar, "Pitsburg Uyku Kalitesi İndeksinin Geçerliği ve Güvenirliği.," Türk Psikiyatr. Derg., vol. 7, no. 2, 1996.
- [Background] Ö. C. Gürkan, "Menopoz semptomları değerlendirme ölçeğinin Türkçe formunun güvenirlik ve geçerliliği.," Hemşirelik Forumu Derg., vol. 3, pp. 30-35, 2005.
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] N. H. ŞAHİN, N. H., Kharbouch, S. B., & Şahin, "Menopozal dönemlerdeki yaşam kalitesinin belirlenmesi.," Florence Nightingale Hemşirelik Dergisi, vol. 15, no. 59, pp. 82-90, 2007.
- [Background] Meehan TC. Therapeutic touch as a nursing intervention. J Adv Nurs. 1998 Jul;28(1):117-25. doi: 10.1046/j.1365-2648.1998.00771.x. PMID 9687138
- [Background] J. Macrae, Therapeutic Touch. izmir: Ege Meta Yayınları, 2000.
- [Derived] Keskin Tore F, Yagmur Y. The effects of therapeutic touch and music on sleep quality, menopausal symptoms, and quality of life in menopausal women. Menopause. 2023 Dec 1;30(12):1221-1229. doi: 10.1097/GME.0000000000002269. Epub 2023 Oct 24. PMID 37874963

DOCUMENTS (3):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT05180266/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT05180266/SAP_001.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT05180266/ICF_002.pdf